CLINICAL TRIAL: NCT02898363
Title: Awareness on Cancer in Persons With Intellectual Disabilities
Acronym: ONCODEFI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AO-INCA/2012/DS-01
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Cancer
Keywords: Care of disabled population; Mental retardation; Cancer screening; Cancer prevention
MeSH Terms: conditions — Neoplasms; Intellectual Disability

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Information campaign — During a two-year information program, physicians, mainly general practitioners, carers in and outside institutions, associations and families will be informed on cancer frequency, on cancer particularities and on cancer detection in persons with intellectual disabilities by means of documents, mails and e-mails, meetings and a website providing all available useful information on cancer in persons with intellectual disabilities.

SUMMARY:
Context People with intellectual disability (PWIDs), nearly 1,300,000 adults and children in France, develop as many cancers as persons in the general population. However, their tumors are different by their particular organ distribution, the age of onset, the biological background (2,000 genetic conditions are associated with an intellectual disability) and above all the unusual clinical presentation. These cancers are not well known from physicians, carers and families, and often discovered late. A recent review of the literature shows many inequalities in the prevention, monitoring, screening, diagnosis and treatment of cancer in these patients. Currently, no population study on clinical features and stage at diagnosis of cancer in PWIDs is available. No interventional research study has been conducted on this subject.

Hypothesis Investigators hypothesize that inequalities in cancer care of PWIDs do not result from a direct link between intellectual disability and cancer, but are related to diagnosis difficulties of these tumors which are not well known, and to difficulties of communication with these patients who do not express easily their symptoms, particularly pain.

DETAILED DESCRIPTION:
The study will first evaluate characteristics of all cancers diagnosed in PWIDs in the department of Hérault (20,000 PWIDs) during the four-year period preceding the intervention. Investigators will cross the data of social network of PWIDs (CREAI Languedoc Roussillon) which covers nearly 90% of PWIDs living in this area, and the Hérault Cancer Registry. Second, during a two-year information program, physicians, mainly general practitioners, carers in and outside institutions, associations and families will be informed on cancer frequency, on cancer particularities and on cancer detection in PWIDs by the mean of documents, mails and e-mails, meetings and a website providing all available useful information on cancer in PWIDs. Third, characteristics of tumors observed during the three years after the beginning of the intervention will be statistically compared to the corresponding tumors before the intervention. This will be done especially for colon cancer and breast cancer using the TNM stage and the used therapeutic means. On the basis of the first part of the study, if a significant difference on stage at diagnosis and treatment is observed compared to the general population, other tumors will also be included in the comparison, if relevant.

ELIGIBILITY:
Inclusion Criteria:

* Persons with intellectual disabilities according to the World Health Organization definition
* Residing in the Hérault department of France
* Diagnosis of a malign invasive or in-situ tumor

Exclusion Criteria:

* Refusal of study participation following provision of information (refusal by the patient, or his/her guardian, or principal caregiver)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is all adults with intellectual disabilities residing in the Hérault department of France who have been diagnosed with cancer
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cancer incidence among persons with intellectual disabilities | Change from baseline (i.e. years -4 through -1) to years 1 through 3

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Satgé, MD, PhD, Study Director — IURC - Laboratoire de Biostatistique d'Epidémiologie et de Recherche Clinique
Locations (1):
- IURC - Laboratoire de Biostatistique d'Epidémiologie et de Recherche Clinique, Montpellier, France